CLINICAL TRIAL: NCT03414476
Title: Demonstration of the Presence of Carbonyl Stress in the Hair Follicles of Women With Reactive Hair Loss
Brief Title: Demonstration of Carbonyl Stress on Hair Follicles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STRESSCARBONYL1
Record Dates: First submitted 2018-01-10; First posted 2018-01-30 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2018-01

CONDITIONS: Effluvium; Telogen

STUDY DESIGN:
Intervention Model Description: 1 group of women with effluvium télogène
  1 group of women without effluvium télogène
Masking Description: Monocentric, Exploratory study, open, comparative, in parallel groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ET group (Experimental): Sampling : Hair follicles sampling on the scalp in women with Telogene Effluvium
  Interventions: Other: Hair follicles sampling
- Control group (Experimental): Sampling: Hair follicles sampling on the scalp in women without Telogene Effluvium
  Interventions: Other: Hair follicles sampling

INTERVENTIONS:
Other: Hair follicles sampling — The follicles will be collected by lock of 10 hair on the scalp (centro-parietal part), to obtain 40 follicles with epithelial sheath

SUMMARY:
In this study, the investigator will try to highlight the presence of carbonyl compounds in the hair follicles of women with telogen effluvium (ET) linked to stress of various origins (fatigue, infectious diseases, emotional stress ...).

DETAILED DESCRIPTION:
At the cutaneous level, oxidative stress induces the formation of carbonyl compounds which, by binding to proteins, produce nonfunctional adducts inducing cutaneous aging. Is this mechanism, called "Carbonyl stress", also present in the scalp and can it be one of the mechanisms involved in the occurrence of reactive hair loss ? To demonstrate this, samples of hair follicles are made. The proteins are extracted from the samples and then assayed. The oxidized (carbonyl) proteins are labeled with specific fluorescent probes.

ELIGIBILITY:
Inclusion Criteria:

Criteria related to the Population :

* Women aged from 18 to 40 ans (included)
* Phototype I à IV included, according to Fitzpatrick Classification
* Hair length 5 cm on the sampling area (centro-parietal part)
* Last shampoo at least 2 days before the inclusion visit, without application of styling product, care or water between this last shampoo and the inclusion
* Informed consent signature

Criteria related to the studied condition:

* ET group: hair loss related to various etiologies evaluated by a questionnaire according to the investigator's opinion and positive pull test (at least 3 hair collected per lock of 50 to 60 hair) AND
* Control group : no hair loss, evaluated by the questionnaire and negative pull test (less than 3 hair collected per lock of 50 to 60 hair)

Exclusion Criteria:

Criteria related to Population :

* Menopause
* Pregnancy, breastfeeding, childbirth for less than 6 months

Criteria related to Pathology :

For both groups:

* Alopecia causing hair loss on the upper part of the scalp
* Dermatological pathology or evolving cutaneous lesion in the scalp
* Control group only:
* Chronic unstabilized condition
* Acute evolving pathology

Criteria related to theTreatments :

For both groups:

* Use for at least 1 month of Minoxidil, Aminexil in the 3 months before inclusion or ongoing
* Systemic treatment affecting hair growth
* Any treatment or dietary supplement for antioxidant or capillary

Control group only:

* Treatment of general thyroid disorders initiated or modified for less than 3 months prior to inclusion
* Treatment of anemia if started less than 3 months before inclusion
* General treatment initiated or modified for less than 3 months prior to inclusion in the study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — women
Enrollment: 40 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2018-06-25 (Actual); Study Completion 2018-06-25 (Actual)

PRIMARY OUTCOMES:
Biological evaluation | Visit 1- Day 1
  Evaluation of the quantity of carbonyl compounds measured in the hair follicles taken from the two groups.

SECONDARY OUTCOMES:
Safety evaluation | Visit 1- Day 1
  Adverse events evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Christine SAINT MARTORY, MD, Principal Investigator — Unaffiliate
Locations (6):
- France (6):
  - Centre hospitalier Lyon Sud, Lyon
  - Centre de Pharmacologie Clinique Appliquée à la Dermatologie, Nice
  - Centre de santé SABOURAUD, Paris
  - INTERTEK France, Paris
  - Centre de Recherche sur la Peau, Toulouse
  - Laboratoire Dermscan, Villeurbanne

IPD SHARING:
Plan to Share IPD: No
Proof of concept study, with confidential data